CLINICAL TRIAL: NCT06564974
Title: Registry Study to Observe Long-term Safety of Vamorolone (AGAMREE®) in Patients With Duchenne Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DMD-001
Record Dates: First submitted 2024-08-09; First posted 2024-08-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Neuromuscular; AGAMREE®
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — VBP15 compound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Vamorolone — Patients on treatment with Vamorolone (AGAMREE®) Dosage: Oral Suspension: 40 mg/mL . Per package insert, the recommended dosage is 6 mg/kg taken orally once daily, up to a maximum daily dosage of 300 mg for patients weighing more than 50 kg.
  Decrease dosage gradually when administered for more than one week.
  Other Names: AGAMREE®

SUMMARY:
The goal of this observational study is to follow patients being treated with the FDA approved drug AGAMREE® in male patients 2 years of age or older with Duchenne's Muscular Dystrophy for long term safety and quality of life.

DETAILED DESCRIPTION:
This is a multi-center, observational, prospective, longitudinal registry designed to collect data in male patients aged 2 years and older with DMD treated with AGAMREE®.

This registry will be conducted in the US, at approximately 25 sites known to treat and follow patients with DMD. The registry plans to enroll approximately 250 male patients aged 2 years and older with DMD.

Evaluations will include:

* Growth parameters
* Body mass index (BMI)
* Vital Signs
* Physical Exam
* Laboratory (Chemistry and Hematology)
* North Star Ambulatory Assessment (NSAA)
* Performance of Upper Limb (PUL)
* Cardiovascular status
* Fractures
* Bone density
* Puberty
* Quality of life (QoL)
* Adverse events (AEs)

Patients will be followed for approximately 5 years in the registry and will return to the site for Yearly Follow-up Visits (+/- 30 days) for registry assessments. Information on standard of care treatment and procedures for management of DMD will also be collected. Patients and/or their parents/legal guardians will be asked to complete paper QoL questionnaires at enrollment and at each Yearly Follow-up Visit (+/- 30 days).

ELIGIBILITY:
Inclusion Criteria:

1. Patient or parent/guardian willing and able to provide written informed consent after the nature of the registry has been explained and before the start of any registry-related procedures.
2. Patient and/or parent/guardian are willing and able to complete QoL questionnaires.
3. Male patients at least 2 years old.
4. Confirmed diagnosis of DMD (via genetic testing or muscle biopsy with absent dystrophin staining to antidystrophin antibodies 3, 1, or 2, or dystrophin immunohistochemistry or western blot).
5. Currently on treatment with AGAMREE®.

Exclusion Criteria:

1. Any contraindication to AGAMREE® or medical condition, which, in the opinion of the investigator, would affect registry participation, performance, or interpretation of registry assessments.

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male subjects 2 years of age and older.
Study Population: Male subjects 2 years of age and older will be selected from DMD centers and Institutions across the US. Subjects will be recruited from the sites respective database.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Change in BMI Z score at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  BMI is in kg/m^2, using Height in CM (centimeters) and Weight in Kgs(kilograms). Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Change in Height Z-score at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  Height is measured in CM (centimeters). Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Change in Puberty development using the Tanner Stage at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  The Tanner Stage measures pubertal development of male external genitalia and pubic hair. This is a uniformly accepted scale and can be conducted by the Investigator or an endocrinologist.
  The scale is 1-5 per the following:
  Male External Genitalia Scale Stage 1: Testicular volume < 4 ml or long axis < 2.5 cm Stage 2: 4 ml-8 ml (or 2.5 to 3.3 cm long), 1st pubertal sign in males Stage 3: 9 ml-12 ml (or 3.4 to 4.0 cm long) Stage 4: 15-20 ml (or 4.1 to 4.5 cm long) Stage 5: > 20 ml (or > 4.5 cm long)
  • Pubic Hair Scale Stage 1: No hair Stage 2: Downy hair Stage 3: Scant terminal hair Stage 4: Terminal hair that fills the entire triangle overlying the pubic region Stage 5: Terminal hair that extends beyond the inguinal crease onto the thigh
  Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Number of Fractures based on Spine x-rays at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  Bone evaluations will be performed through lateral spine x-ray, Anteroposterior (AP) spine x-ray, and dual-energy x-ray absorptiometry.
Presence or absence of Cataracts at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  Cataracts will be assessed by an ophthalmologist based on a Comprehensive Eye Exam to include the Slit Lamp test.
Presence of Cardiomyopathy at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  Cardiomyopathy will be assessed by echocardiography using transmural strain profile (TMSP) analysis.
Evaluation of Hormonal status based on Cortisol levels at enrollment. | At enrollment
  Morning cortisol ( before 10 AM) levels will be measured in ug/dl by a Central Lab. The normal range is 3.7-19.4 ug/dl.
Presence or absence of Glaucoma at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  Glaucoma will be assessed by an ophthalmologist based on a Comprehensive Eye Exam and testing intraocular pressure.
Number of patients experiencing any Adverse Events (AEs) or Serious Adverse Events (SAEs) after signing the Informed Consent Form. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  Adverse Events (AEs)/ Serious Adverse Events (SAEs) will be assessed by the current version of the CTCAE at the time the adverse event is identified, and will be summarized by MedDRA system organ class and preferred term using the current version of MedDRA.
Change in Pediatric Quality of Life Inventory Duchenne Muscular Dystrophy (PedsQL DMD) Module at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  PedsQL DMD is self-reported. It consists of 18 items in 4 domains. Daily Activities' (5 items),Treatment' (4 items), 'Worry' (6 items) and 'Communication' (3 items). 5-point response scale to indicate how much of a problem each item has been in the past month (0 = never a problem to 4 = almost always a problem). Items are reverse scored and linearly transformed to a 0-100 scale, so that higher scores indicate better QoL.
  Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Change in Duchenne Muscular Dystrophy Quality of Life (DMD-QoL)at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  The DMD-QoL is a 14-item questionnaire. The questionnaire is answered using a 4-point response scale (Never, Sometimes, A lot of the time, All of the time). The DMD-QoL has a hierarchical (or 'higher-order') factor structure, with 3 lower-order factors (physical, social, and psychological) and 1 higher-order factor (overall QoL, comprised of the 3 lower-order factors). Higher scores represent a more positive QoL (overall or within each subscale).
  Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Change in Euro Qol 5 Dimensions (EQ-5D) at the End-of-Registry ( 5 years) or Early-Termination. | t enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  The EQ-5D-5L (5-Levels) will be completed by patients aged 16 years and older or Parent/guardian. The EQ-5D-5L consists of a descriptive system of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and 5 levels (1, no problems; 2, slight problems; 3, moderate problems; 4, severe problems; 5, extreme problems), and a visual analog scale (VAS) from 0 (worst health) to 100 (best health). Patients aged 8 to 15 years will complete the EQ-5D-Y-3L (Youth) questionnaire. The EQ-5D-Y-3L consists of a descriptive system of 5 dimensions and 3 levels (no problems, some problems, and a lot of problems), and a visual analog scale. Parents/legal guardian of patients aged 4 to 7 years will complete the EQ-5D-Y-3L proxy version, which rates how the parent/legally authorized representative rates the health of the child.
  Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Change in Patient Reported Outcome Measure for the Upper Limb (PROM UL) at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  The PROM UL consists of 32 items covering four domains of activities of daily living: (1) food, (7 items, max score 14); (2) self-care, (8 items, max score 16); (3) household and environment, (6 items, max score 12); (4) leisure and communication, (11 items, max score 22). For each question, the patients and/or their parents/legal guardian are asked to report their perceived difficulty in performing the activity on a 3-level scale: Cannot do (0); Can do with difficulty (1); Can do easily (2). The maximum total score is 64.
  Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Change in North Star Ambulatory Assessment (NSAA) at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  The NSAA is a clinical assessment scale specifically designed to measure functional ability in ambulant male patients. The NSAA consists of 17 scored items and 2 timed tests, including the Time to Run/Walk Test (TTRW) and the Time to Stand Test (TTSTAND).
  The TTRW measures the time (in seconds) that it takes the patient to run or walk 10 meters.
  The TTSTAND measures the time (in seconds) required for the patient to stand in an erect position from supine (floor).
  Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.
Change in Performance of Upper Limb (PUL) at the End-of-Registry ( 5 years) or Early-Termination. | At enrollment, at each Yearly Follow-up Visit (+/- 30 days), and at the End-of-Registry ( 5 years) or Early-Termination.
  The PUL module is a tool designed for assessing upper limb function in ambulant and non-ambulant patients. The PUL module consists of 22 items with an entry item to define the starting functional level (which corresponds to the Brooke scale) and 21 items subdivided into shoulder level (4 items), elbow level (9 items), and distal (i.e., wrist and fingers) level (8 items). For weaker patients, a low score on the entry item (i.e., less than 4 points) means that shoulder-level items do not need to be performed. Each dimension can be scored separately with a maximum score of 16 for the shoulder level, 34 for the elbow level, and 24 for the distal level. A total score can be achieved by adding the three-level scores, with a maximum global score of 74 points.
  Change = End-of Registry ( 5 Years) or (early enrollment termination) minus (-) Enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: William Andrews, MD, Study Director — Catalyst Pharmaceuticals; Aravindham Veerapandiyan, MD, Principal Investigator — Arkansas Childrens Hospital
Locations (25):
- United States (23):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - University of Florida Clinical and Translational Science Institue, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University Health - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Massachusetts Memorial Medical Center, North Worcester, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Atrium Health Neurosciences Institute, Charlotte, North Carolina
  - Duke University Medical Center and Childrens Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center- Penn State Hershey Neuroscience Institute, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Neurology Rare Disease Center - Neurology & Neuromuscular Care Center, Denton, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Health System (UVAHS) - Pediatric Neuromuscular Center, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan, Puerto Rico
  - FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No